CLINICAL TRIAL: NCT03452137
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of Atezolizumab (Anti-PD-L1 Antibody) as Adjuvant Therapy After Definitive Local Therapy in Patients With High-Risk Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: A Study of Atezolizumab (Anti-PD-L1 Antibody) as Adjuvant Therapy After Definitive Local Therapy in Patients With High-Risk Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Acronym: IMvoke010
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision to terminate the study as its primary endpoint of investigator-assessed event free survival (INV-EFS) was not met at its final EFS analysis. No new safety signals were identified.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WO40242; 2017-003302-40 (EudraCT Number)
Record Dates: First submitted 2018-02-25; First posted 2018-03-02 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Locally Advanced Squamous Cell Carcinoma of the Head and Neck (SCCHN)
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezolizumab (Active Comparator): Participants will receive Atezolizumab for 16 cycles, or up to 1 year (whichever occurs first)
  Interventions: Drug: Atezolizumab
- Placebo (Experimental): Participants will receive Placebo for 16 cycles, or up to 1 year (whichever occurs first).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab intravenous infusion will be administered at a fixed dose on Day 1 of each 21-day cycle for 16 cycles.
  Arms: Atezolizumab
Drug: Placebo — Placebo intravenous infusion will be administered a fixed dose on Day 1 of each 21-day cycle for 16 cycles.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of atezolizumab compared with placebo as adjuvant therapy after definitive local therapy in patients with high-risk locally advanced squamous cell carcinoma of the head and neck (SCCHN)

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed Squamous Cell Carcinoma of the Head and Neck (SCCHN)
* Human Papilloma Virus (HPV) status
* Completed definitive local therapy
* Absence of metastatic disease as documented by radiographic scans
* Adequate hematologic and end-organ function
* For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
* For women of childbearing potential: agreement to remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 5 months after the last dose of study treatment. Women must refrain from donating eggs during this same period.
* Confirmed response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) to definitive local therapy documented by CT with contrast or MRI with contract to head and neck region done >= 8 weeks after completion of definitive local therapy and within 28 days prior to initiation of study drug.

Exclusion Criteria:

* Patients who have received surgery alone or radiotherapy alone as definitive local therapy
* Squamous cell carcinoma of the nasopharynx or paranasal sinuses or non-squamous histology
* Evidence of disease progression or metastatic disease during or following definitive local therapy documented in post-definitive local therapy screening scans
* Uncontrolled or symptomatic hypercalcemia
* Active or history of autoimmune disease or immune deficiency
* Active tuberculosis
* Significant cardiovascular disease
* History of malignancy, including prior SCCHN primary tumors within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Prior allogeneic stem cell or solid organ transplantation
* Current treatment with anti-viral therapy for Hepatitis B Virus (HBV)
* Treatment with systemic immunostimulatory agents
* Treatment with systemic immunosuppressive medication
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the last dose of study treatment
* Patients who have received a non-FDA or non-EMA approved anti-EGFR agent or any other non-FDA or non-EMA, approved agent as part of definitive local therapy, unless the unapproved agent was given in addition to an approved agent
* Any systemic therapies after permitted definitive local therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2024-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (135):
- United States (12):
  - City of Hope National Medical Center, Duarte, California
  - University of California San Diego Medical Center; Moores Cancer Center, La Jolla, California
  - UCLA Hematology/Oncology, Santa Monica, California
  - Miami Cancer Institute of Baptist Health, Inc., Miami, Florida
  - Woodlands Medical Specialists, P.A., Pensacola, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, a Service of WellStar Cobb Hospital, Marietta, Georgia
  - Cancer Center of Kansas, Wichita, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Billings Clinic Research Center, Billings, Montana
  - Cleveland Clinic; Taussig Cancer Institute, Cleveland, Ohio
  - Blue Ridge Cancer Care, Roanoke, Virginia
- Australia (4):
  - St George Hospital, Kogarah, New South Wales
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Peter MacCallum Cancer Center, North Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Clinique Ste-Elisabeth, Namur, Belgium
- Brazil (7):
  - Santa Casa de Misericordia de Salvador, Salvador, Estado de Bahia
  - Hospital do Cancer de Pernambuco - HCP, Recife, Pernambuco
  - Instituto Nacional de Cancer - INCa; Oncologia, Rio de Janeiro, Rio de Janeiro
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina do ABC - FMABC, Santo André, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario
- China (9):
  - Beijing Cancer Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai East Hospital, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Zhejiang Cancer Hospital, Zhejiang
- France (9):
  - Institut Sainte Catherine, Avignon
  - Centre Georges Francois Leclerc, Dijon
  - CENTRE LEON BERARD; Département d?Hématologie et d?Oncologie, Lyon
  - Hopital Timone Adultes; Oncologie Medicale Et Usp, Marseille
  - ICM; Radiotherapie, Montpellier
  - Hopital Tenon; Oncologie Radiotherapie, Paris
  - CHU Bordeaux, Pessac
  - Hôpitaux D'Instruction Des Armees Begin, Saint-Mandé
  - Gustave Roussy Cancer Campus; Radiotherapie, Villejuif
- Germany (4):
  - Universitätsklinikum Bonn; Med. Klinik und Poliklinik III; Hämatologie, Onkologie und Rheumatologie, Bonn
  - Universitätsklinikum Freiburg, Klinik für Strahlenheilkunde, Freiburg im Breisgau
  - Klinikum d. Uni. München; Campus Großhadern; Klinik und Poliklinik f. Strahlenthera. und Radioonko, München
  - Universitätsmedizin Rostock, Klinik und Poliklinik für Strahlentherapie; Zentrum für Radiologie, Rostock
- Hungary (3):
  - Orszagos Onkologial Intezet; Onkologiai Osztaly X, Budapest
  - Budapesti Uzsoki Utcai Kórház, Budapest
  - Pécsi Tudományegyetem; Klinikai Központ Onkoterápiás Intézet, Pécs
- India (2):
  - Medanta-The Medicity, Gurgaon, Haryana
  - Tata Memorial Hospital; Dept of Medical Oncology, Mumbai, Maharashtra
- Italy (11):
  - Istituto Nazionale Tumori Fondazione G. Pascale; S.C. Oncol. Medica Testa-Collo e Sarcoma, Napoli, Campania
  - Ospedale Umberto I ASL di Ravenna Presidio Ospedaliero di Lugo, Lugo, Emilia-Romagna
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - Policlinico Umberto i di Roma; dip. Scienze Radiologiche, Oncologiche, Anatomopatologiche, Rome, Lazio
  - Ospedale Civile; Servizio Oncologia, Savona, Liguria
  - Spedali Civili di Brescia, Brescia, Lombardy
  - Fondazione IRCCS Istituto Nazionale dei Tumori;S.S. Trattamento MedicoTumori dellaTesta e delCollo, Milan, Lombardy
  - Asst Santi Paolo E Carlo; Unita Operativa Di Oncologia Medica, Milan, Lombardy
  - Istituto Clinico Humanitas;U.O. Oncologia Medica Ed Ematologia, Rozzano, Lombardy
  - Azienda Ospedaliero-Universitaria Careggi; SOD Radioterapia, Florence, Tuscany
  - IOV - Istituto Oncologico Veneto IRCCS, Padua, Veneto
- Japan (14):
  - Aichi Cancer Center Hospital, Aichi
  - National Cancer Center Hospital East, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hokkaido University Hospital, Hokkaido
  - Kobe University Hospital, Hyōgo
  - Miyagi Cancer Center, Miyagi
  - Okayama University Hospital, Okayama
  - Osaka International Cancer Institute, Osaka
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - The Jikei University Hospital, Tokyo
  - Tokyo Medical and Dental University Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Tokyo Medical University Hospital, Tokyo
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne; Klinika Onkologii i Radioterapii, Gdansk
  - Narodowy Inst.Onkol.im.Sklodowskiej-Curie Panstw.Inst.Bad Gliwice; III Klin. Radioter. i Chemioter., Gliwice
  - Narodowy Inst.Onkologii im.Sklodowskiej-Curie Panstw.Inst.Bad; Klinika Nowotworów G?owy i Szyi, Warsaw
- Portugal (3):
  - IPO de Coimbra; Servico de Oncologia Medica, Coimbra
  - Hospital de Santa Maria; Servico de Oncologia Medica, Lisbon
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Russia (11):
  - Krasnoyarsk Regional Oncology Dispensary n.a. Krizhanovsky; Chemotherapy, Krasnoyarsk, Krasnodarskiy Kray
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - Main Military Clinical Hospital named after N.N. Burdenko, Moscow, Moscow Oblast
  - P.A. Herzen Oncological Inst. ; Oncology, Moscow, Moscow Oblast
  - First MSMU n.a. Sechenov Univercity Hospital 1; Plastic surgery, Moskva, Moscow Oblast
  - FSAI Treatment and rehabilitation Centre Ministry of Health; Clinical research and chemotherapy., Moskva, Moscow Oblast
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg, Sankt-Peterburg
  - Sverdlovsk Regional Oncology Dispensary; Chemotherapy, Yekaterinburg, Sverdlovsk Oblast
  - Novosibirsk Regional Oncological Dispancer, Novosibirsk
  - BHI of Omsk region Clinical Oncology Dispensary, Omsk
  - Tomsk scientific research institute of oncology SO RAMN, PAD; Pathological, Tomsk
- South Africa (4):
  - Tygerberg Hospital; Oncology Dept, Cape Town
  - GVI Oncology Outeniqua Unit, George
  - The Oncology Centre; Haematology - Radiation Oncology, Mayville
  - Steve Biko Academic Hospital; Oncology, Pretoria
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Badalona, Barcelona
  - Insititut Catala D'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario de Salamanca; Servicio de Oncologia, Salamanca
  - Hospital Univ. Nuestra Señora de Valme; Servicio de Oncologia, Seville
  - Hospital Universitario la Fe; Servicio de Oncologia, Valencia
- Taiwan (5):
  - China Medical University Hospital;Oncology and Hematology Office Critical Care Center, 14H, Taichung
  - Taichung Veterans General Hospital; Radiation Oncology, Taichung
  - National Cheng Kung University Hospital; Oncology, Tainan
  - Division of Hematology and Oncology, Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital; Oncology, Zhongzheng Dist.
- Thailand (3):
  - Ramathibodi Hospital; Dept of Med.-Div. of Med. Onc, Bangkok
  - Faculty of Med. Siriraj Hosp.; Med.-Div. of Med. Oncology, Bangkok
  - Songklanagarind Hospital; Department of Oncology, Songkhla
- Turkey (Türkiye) (4):
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Dr. Abdurrahman Yurtarslan Oncology Hospital; 2nd Oncology Clinic, Ankara
  - Gazi University Medical Faculty, Oncology Hospital, Ankara
  - ?zmir Medical Point; Oncology, Kar?iyaka
- Ukraine (7):
  - Municipal Noncommercial Institution Regional Center of Oncology, Kharkiv, Kharkiv Governorate
  - Vinnytsya Regional Clinical Oncology Dispensary, Vinnytsia, Podolia Governorate
  - Ivano-Frankivsk Regional Oncology Center, Ivano-Frankivsk
  - Kyiv City Clinical Oncological Center, Day Hospital Department for Oncological patients, Kiev
  - ME Kryviy Rih Oncology Dispensary of Dnipropetrovs?k Regional Council; Chemotherapy Department, Kryvyi Rih
  - Lviv State Oncology Regional Treatment and Diagnostic Centre; Department of hemotherapy, Lviv
  - RCI Sumy Regional Clinical Oncological Dispensary, Sumy
- United Kingdom (5):
  - Aberdeen Royal Infirmary; Medical Oncology Dept, Aberdeen
  - Velindre Cancer Centre, Cardiff
  - The Royal Marsden Hospital, Fulham, London
  - Derriford Hospital, Plymouth
  - Royal Marsden NHS Foundation Trust, Sutton

REFERENCES:
- [Derived] Haddad R, Fayette J, Teixeira M, Prabhash K, Mesia R, Kawecki A, Dechaphunkul A, Dinis J, Guo Y, Masuda M, Hsieh CY, Ghi MG, Vaz de Melo Sette C, Harrington K, Tahara M, Saba NF, Lau A, Jiang T, Yan Y, Ballinger M, Kaul M, Matheny C, Cuchelkar V, Wong DJ. Atezolizumab in High-Risk Locally Advanced Squamous Cell Carcinoma of the Head and Neck: A Randomized Clinical Trial. JAMA. 2025 May 13;333(18):1599-1607. doi: 10.1001/jama.2025.1483. PMID 40079944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study across 128 investigative sites in 23 countries from 03 April 2018 to 06 March 2024.
Pre-assignment Details: A total of 406 participants with locally advanced squamous cell carcinoma of the head and neck (SCCHN) were randomized in 1:1 ratio to receive either atezolizumab or placebo.
Groups:
- Placebo: Participants received atezolizumab matching placebo, intravenous (IV) infusion on Day 1 of each 21-day cycle for 16 cycles or up to 1 year or until disease recurrence, disease progression, unacceptable toxicity, consent withdrawal, or study termination by sponsor, whichever occurred first.
- Atezolizumab: Participants received atezolizumab 1200 milligrams (mg), IV infusion on Day 1 of each 21-day cycle for 16 cycles or up to 1 year or until disease recurrence, disease progression, unacceptable toxicity, consent withdrawal, or study termination by sponsor, whichever occurred first.
Period: Overall Study
Arm/Group | Placebo | Atezolizumab
Started | 203 | 203
Received at Least One Dose of Study Drug (Safety-Evaluable Population) | 203 | 202
Completed | 0 | 0
Not Completed | 203 | 203
Not completed — Death | 67 | 70
Not completed — Lost to Follow-up | 4 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Study Terminated by Sponsor | 120 | 121
Not completed — Withdrawal by Subject | 12 | 9

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants, regardless of whether they received any of the assigned treatment.
Groups:
- Placebo: Participants received atezolizumab matching placebo, IV infusion on Day 1 of each 21-day cycle for 16 cycles or up to 1 year or until disease recurrence, disease progression, unacceptable toxicity, consent withdrawal, or study termination by sponsor, whichever occurred first.
- Atezolizumab: Participants received atezolizumab 1200 mg, IV infusion on Day 1 of each 21-day cycle for 16 cycles or up to 1 year or until disease recurrence, disease progression, unacceptable toxicity, consent withdrawal, or study termination by sponsor, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Placebo | Atezolizumab | Total
Number analyzed (Participants) | 203 | 203 | 406
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (10.1) | 59.4 (8.5) | 58.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 35 | 64
  Male | 174 | 168 | 342
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 11 | 24
  Not Hispanic or Latino | 181 | 183 | 364
  Unknown or Not Reported | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 61 | 68 | 129
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 135 | 121 | 256
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 12 | 18
Human papilloma virus (HPV) Status [Count of Participants; unit: Participants]
  Negative | 166 | 168 | 334
  Positive | 37 | 35 | 72
Type of Definitive Local Therapy [Count of Participants; unit: Participants]
  Primary Surgery | 78 | 79 | 157
  No Primary Surgery | 125 | 124 | 249
Response to Definitive Local Therapy [Count of Participants; unit: Participants] — Responses were assessed according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1).
  Participants
    Complete Response (CR) | 170 | 170 | 340
    Partial Response (PR) or Stable Disease (SD) | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Investigator-Assessed Event-Free Survival (INV-assessed EFS)
Description: EFS was defined as the time from randomization to the first documented disease recurrence (per unequivocal radiographic evidence of local recurrence, new second primary SCCHN lesion, or development of distant metastasis), or disease progression [per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)] per assessment by investigator, or death from any cause, whichever occurred first. Progressive disease (PD) was defined as at least a 20% increase in the sum of diameters (SOD) of target lesions, taking as reference the smallest SOD on study (including baseline). Participants without disease recurrence, progression or death at the time of analysis were censored at the time of the last tumor assessment. EFS was estimated using the Kaplan-Meier method.
Time Frame: Randomization to the first documented disease recurrence, disease progression or death from any cause, whichever occurs first (up to 5 years)
Population: ITT population included all randomized participants, regardless of whether they received any of the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Atezolizumab
Number analyzed (Participants) | 203 | 203
months | 52.73 [41.43 to NA] — The upper limit of the 95% confidence interval (CI) was not estimable for INV-EFS because there was an insufficient number of events. | 59.47 [46.75 to NA] — The upper limit of the 95% CI was not estimable for INV-EFS because because there was an insufficient number of events.
Statistical Analysis 1: Comparison: Placebo vs Atezolizumab; Stratified Analysis: The stratification factors were response to definitive local therapy, human papillomavirus (HPV) status and type of definitive local therapy as per interactive voice or web-based response system (IxRS); Test type: Superiority; p = 0.6804, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.70 to 1.26] — HR was estimated by Cox regression

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause. Data from participants who were alive at the time of the analysis was censored as of the last date they were known to be alive. OS was estimated using the Kaplan-Meier method.
Time Frame: Randomization to death from any cause (up to 5 years, 5 months)
Population: ITT population included all randomized participants, regardless of whether they received any of the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Atezolizumab
Number analyzed (Participants) | 203 | 203
months | NA [NA to NA] — The median and lower and upper limits of the 95% CI for OS were not estimable because there was an insufficient number of events. | NA [59.47 to NA] — The median and upper limit of the 95% CI for OS were not estimable because there was an insufficient number of events.
Statistical Analysis 1: Comparison: Placebo vs Atezolizumab; Stratified Analysis: The stratification factors were response to definitive local therapy, HPV status and type of definitive local therapy as per interactive voice or web-based response system (IxRS); Test type: Superiority; p = 0.8371, Log Rank; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.68 to 1.36] — HR was estimated by Cox regression

3. Secondary Outcome: Independent Review Facility (IRF) Assessed EFS
Description: EFS was defined as the time from randomization to the first documented disease recurrence (per unequivocal radiographic evidence of local recurrence, new second primary SCCHN lesion, or development of distant metastasis), or disease progression (per RECIST v1.1) per assessment by IRF, or death from any cause, whichever occurred first. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD on study (including baseline). Participants without disease recurrence, progression or death at the time of analysis were censored at the time of the last tumor assessment. EFS was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: ITT population included all randomized participants, regardless of whether they received any of the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Atezolizumab
Number analyzed (Participants) | 203 | 203
months | 52.73 [43.10 to NA] — The upper limit of the 95% CI was not estimable for IRF-EFS because there was an insufficient number of events. | 59.47 [45.17 to NA] — The upper limit of the 95% CI was not estimable for IRF-EFS because there was an insufficient number of events.
Statistical Analysis 1: Comparison: Placebo vs Atezolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.9115, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.73 to 1.32] — HR was estimated by Cox regression

4. Secondary Outcome: Percentage of Participants Event-Free for IRF-assessed EFS at 1, 2, 3, and 4 Years
Description: EFS was defined as the time from randomization to the first documented disease recurrence (per unequivocal radiographic evidence of local recurrence, new second primary SCCHN lesion, or development of distant metastasis), or disease progression (per RECIST v1.1) per assessment by IRF, or death from any cause, whichever occurred first. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD on study (including baseline). Participants without disease recurrence, progression or death at the time of analysis were censored at the time of the last tumor assessment. Kaplan-Meier approach was used to estimate percentage of participants who were event-free for EFS at 1, 2, 3 & 4 years.
Time Frame: From randomization to EFS event or date last known to be alive and event-free at 1, 2, 3, and 4 years
Population: ITT population included all randomized participants, regardless of whether they received any of the assigned treatment. Number analyzed per timepoint are unique number of participants out of all the assessed participants who remain at risk for an EFS event at that timepoint. Different participants may have contributed data for each timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Atezolizumab
Number analyzed (Participants) | 203 | 203
percentage of participants
  1 Year: number analyzed (Participants) | 143 | 142
  1 Year | 72.59 [66.41 to 78.77] | 71.92 [65.68 to 78.16]
  2 Year: number analyzed (Participants) | 124 | 128
  2 Year | 65.85 [59.25 to 72.46] | 66.31 [59.73 to 72.89]
  3 Year: number analyzed (Participants) | 108 | 115
  3 Year | 59.87 [52.99 to 66.76] | 61.07 [54.25 to 67.88]
  4 Year: number analyzed (Participants) | 63 | 66
  4 Year | 54.71 [47.51 to 61.90] | 54.72 [47.52 to 61.91]
Statistical Analysis 1: Comparison: Placebo vs Atezolizumab; Difference in EFS Event-Free Rates at 1 year; Test type: Superiority; p = 0.8816, Z test; Difference in Event Free Rate = -0.67, 95% CI 2-sided [-9.45 to 8.11]
Statistical Analysis 2: Comparison: Placebo vs Atezolizumab; Difference in EFS Event-Free Rates at 2 years; Test type: Superiority; p = 0.9234, Z test; Difference in Event Free Rate = 0.46, 95% CI 2-sided [-8.86 to 9.78]
Statistical Analysis 3: Comparison: Placebo vs Atezolizumab; Difference in EFS Event-Free Rates at 3 years; Test type: Superiority; p = 0.8090, Z test; Difference in Event Free Rate = 1.19, 95% CI 2-sided [-8.49 to 10.88]
Statistical Analysis 4: Comparison: Placebo vs Atezolizumab; Difference in EFS Event-Free Rates at 4 years; Test type: Superiority; p = 0.9985, Z test; Difference in Event Free Rate = 0.01, 95% CI 2-sided [-10.17 to 10.19]

5. Secondary Outcome: Percentage of Participants Event-Free for INV-assessed EFS at 1, 2, 3, and 4 Years
Description: EFS was defined as the time from randomization to the first documented disease recurrence (per unequivocal radiographic evidence of local recurrence, new second primary SCCHN lesion, or development of distant metastasis), or disease progression (per RECIST v1.1) per assessment by the investigator, or death from any cause, whichever occurred first. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD on study (including baseline). Participants without disease recurrence, progression or death at the time of analysis were censored at the time of the last tumor assessment. Kaplan-Meier approach was used to estimate percentage of participants who were event-free for EFS at 1, 2, 3 & 4 years.
Time Frame: From randomization to EFS event or date last known to be alive and event-free at 1, 2, 3, and 4 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Atezolizumab
Number analyzed (Participants) | 203 | 203
percentage of participants
  1 Year: number analyzed (Participants) | 143 | 151
  1 Year | 70.84 [64.58 to 77.10] | 76.01 [70.09 to 81.93]
  2 Year: number analyzed (Participants) | 124 | 131
  2 Year | 63.81 [57.17 to 70.45] | 67.41 [60.90 to 73.92]
  3 Year: number analyzed (Participants) | 110 | 118
  3 Year | 58.57 [51.73 to 65.41] | 61.71 [54.94 to 68.49]
  4 Year: number analyzed (Participants) | 64 | 70
  4 Year | 55.51 [48.49 to 62.52] | 56.82 [49.75 to 63.88]
Statistical Analysis 1: Comparison: Placebo vs Atezolizumab; Difference in EFS Event-Free Rates at 1 year; Test type: Superiority; p = 0.2393, Z test; Difference in Event Free Rate = 5.17, 95% CI 2-sided [-3.44 to 13.79]
Statistical Analysis 2: Comparison: Placebo vs Atezolizumab; Difference in EFS Event-Free Rates at 2 years; Test type: Superiority; p = 0.4472, Z test; Difference in Event Free Rate = 3.61, 95% CI 2-sided [-5.69 to 12.90]
Statistical Analysis 3: Comparison: Placebo vs Atezolizumab; Difference in EFS Event-Free Rates at 3 years; Test type: Superiority; p = 0.5222, Z test; Difference in Event Free Rate = 3.14, 95% CI 2-sided [-6.49 to 12.77]
Statistical Analysis 4: Comparison: Placebo vs Atezolizumab; Difference in EFS Event-Free Rates at 4 years; Test type: Superiority; p = 0.7967, Z test; Difference in Event Free Rate = 1.31, 95% CI 2-sided [-8.64 to 11.26]

6. Secondary Outcome: Percentage of Participants Event-Free for OS at 2, 3, and 5 Years
Description: OS was defined as the time from randomization to death from any cause. Data from participants who were alive at the time of the analysis was censored as of the last date they were known to be alive. Kaplan-Meier approach was used to estimate the percentage of participants who were event-free for OS at 2, 3 and 5 years.
Time Frame: From randomization to OS event or date last known to be alive at 2, 3, and 5 Years
Population: ITT population included all randomized participants, regardless of whether they received any of the assigned treatment. Number analyzed per timepoint are unique number of participants out of all the assessed participants who remain at risk for an OS event at that timepoint. Different participants may have contributed data for each timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Atezolizumab
Number analyzed (Participants) | 203 | 203
percentage of participants
  2 Year: number analyzed (Participants) | 157 | 163
  2 Year | 79.23 [73.64 to 84.82] | 82.00 [76.68 to 87.33]
  3 Year: number analyzed (Participants) | 143 | 140
  3 Year | 73.59 [67.48 to 79.70] | 72.34 [66.11 to 78.56]
  5 Year: number analyzed (Participants) | 6 | 6
  5 Year | 62.00 [53.46 to 70.55] | 60.93 [48.01 to 73.86]
Statistical Analysis 1: Comparison: Placebo vs Atezolizumab; Difference in OS Event-Free Rates at 2 years; Test type: Superiority; p = 0.4819, Z test; Difference in Event Free Rate = 2.77, 95% CI 2-sided [-4.95 to 10.49]
Statistical Analysis 2: Comparison: Placebo vs Atezolizumab; Difference in OS Event-Free Rates at 3 years; Test type: Superiority; p = 0.7783, Z test; Difference in Event Free Rate = -1.25, 95% CI 2-sided [-9.97 to 7.47]
Statistical Analysis 3: Comparison: Placebo vs Atezolizumab; Difference in OS Event-Free Rates at 5 years; Test type: Superiority; p = 0.8924, Z test; Difference in Event Free Rate = -1.07, 95% CI 2-sided [-16.56 to 14.42]

7. Secondary Outcome: Change From Baseline in Physical Function (PF) as Assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire- Core 30 (EORTC-QLQ-C30) Score
Description: EORTC QLQ-C30 scale consists of 30 questions that assess participant functioning (physical, emotional, role, cognitive, and social), symptoms (fatigue, nausea and vomiting, pain), global health/quality of life (QoL), and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Change in PF was assessed using the PF scale, where participant responses to 5 questions about daily activities (strenuous activities, long walks, short walks, bed/chair rest & needing help with eating, dressing, washing themselves, or using the toilet) was scored on a 4-point scale (1=Not at All to 4=Very Much). Scores were linearly transformed on a scale of 0 to 100, with a high score indicating worst functioning.
Time Frame: Baseline, Day 1 of Cycles 2 to 16 (Cycle length = 21 days); study discontinuation visit (up to 1 year); Follow-up approximately every 3 months until disease recurrence or progression (up to approximately 4.5 years)
Population: ITT population included all randomized participants, regardless of whether they received any of the assigned treatment. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Atezolizumab
Number analyzed (Participants) | 201 | 200
score on a scale
  Baseline (Cycle 1 Day 1) | 82.78 (16.36) | 83.46 (16.79)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 195 | 193
  Change at Cycle 2 Day 1 | 2.40 (11.09) | -0.58 (10.54)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 194 | 186
  Change at Cycle 3 Day 1 | 3.75 (12.03) | -0.13 (12.62)
  Change at Cycle 4 Day 1: number analyzed (Participants) | 177 | 179
  Change at Cycle 4 Day 1 | 2.90 (13.00) | 0.77 (13.42)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 171 | 168
  Change at Cycle 5 Day 1 | 4.69 (13.86) | 1.60 (12.15)
  Change at Cycle 6 Day 1: number analyzed (Participants) | 169 | 162
  Change at Cycle 6 Day 1 | 4.03 (12.76) | 2.18 (13.87)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 162 | 154
  Change at Cycle 7 Day 1 | 4.33 (13.07) | 3.56 (13.68)
  Change at Cycle 8 Day 1: number analyzed (Participants) | 156 | 151
  Change at Cycle 8 Day 1 | 4.63 (13.07) | 3.19 (13.71)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 152 | 147
  Change at Cycle 9 Day 1 | 4.62 (13.86) | 2.96 (14.41)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 148 | 143
  Change at Cycle 10 Day 1 | 4.41 (14.30) | 2.12 (14.22)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 145 | 139
  Change at Cycle 11 Day 1 | 3.82 (14.20) | 3.69 (12.43)
  Change at Cycle 12 Day 1: number analyzed (Participants) | 143 | 139
  Change at Cycle 12 Day 1 | 4.35 (15.23) | 3.05 (14.89)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 138 | 136
  Change at Cycle 13 Day 1 | 5.62 (13.63) | 3.30 (15.02)
  Change at Cycle 14 Day 1: number analyzed (Participants) | 134 | 129
  Change at Cycle 14 Day 1 | 6.73 (13.67) | 3.20 (13.36)
  Change at Cycle 15 Day 1: number analyzed (Participants) | 133 | 124
  Change at Cycle 15 Day 1 | 6.13 (13.11) | 3.99 (12.92)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 122 | 116
  Change at Cycle 16 Day 1 | 5.92 (14.85) | 4.11 (12.88)
  Change at Study Discontinuation: number analyzed (Participants) | 181 | 175
  Change at Study Discontinuation | 2.94 (16.52) | 2.70 (14.20)
  Change at Follow Up 1: number analyzed (Participants) | 51 | 50
  Change at Follow Up 1 | 1.47 (16.36) | -6.63 (24.41)
  Change at Follow Up 2: number analyzed (Participants) | 42 | 44
  Change at Follow Up 2 | -1.15 (18.10) | 0.19 (17.34)
  Change at Follow Up 3: number analyzed (Participants) | 35 | 33
  Change at Follow Up 3 | -0.81 (17.17) | 2.68 (18.75)
  Change at Follow Up 4: number analyzed (Participants) | 36 | 28
  Change at Follow Up 4 | -1.90 (18.62) | -2.56 (28.57)
  Change at Follow Up 5: number analyzed (Participants) | 30 | 21
  Change at Follow Up 5 | -2.00 (26.21) | -6.03 (35.58)
  Change at Follow Up 6: number analyzed (Participants) | 30 | 18
  Change at Follow Up 6 | -3.61 (18.08) | -3.24 (23.84)
  Change at Follow Up 7: number analyzed (Participants) | 20 | 13
  Change at Follow Up 7 | -6.75 (21.85) | 1.54 (24.82)
  Change at Follow Up 8: number analyzed (Participants) | 20 | 11
  Change at Follow Up 8 | -13.08 (28.96) | 1.36 (33.11)
  Change at Follow Up 9: number analyzed (Participants) | 11 | 9
  Change at Follow Up 9 | 2.88 (14.38) | 4.63 (17.36)
  Change at Follow Up 10: number analyzed (Participants) | 7 | 8
  Change at Follow Up 10 | -16.43 (32.50) | 3.33 (13.80)
  Change at Follow Up 11: number analyzed (Participants) | 10 | 4
  Change at Follow Up 11 | -10.00 (35.31) | -16.67 (24.65)
  Change at Follow Up 12: number analyzed (Participants) | 6 | 4
  Change at Follow Up 12 | -6.67 (8.43) | 0.00 (14.40)
  Change at Follow Up 13: number analyzed (Participants) | 7 | 3
  Change at Follow Up 13 | -5.71 (7.13) | 4.44 (10.18)
  Change at Follow Up 14: number analyzed (Participants) | 3 | 1
  Change at Follow Up 14 | -17.78 (42.86) | -6.67 (0)
  Change at Follow Up 15: number analyzed (Participants) | 4 | 0
  Change at Follow Up 15 | -5.00 (6.38) |
  Change at Follow Up 16: number analyzed (Participants) | 3 | 0
  Change at Follow Up 16 | 2.22 (10.18) |
  Change at Follow Up 17: number analyzed (Participants) | 2 | 0
  Change at Follow Up 17 | -3.33 (4.71) |
  Change at Follow Up 18: number analyzed (Participants) | 2 | 0
  Change at Follow Up 18 | 13.33 (0) |

8. Secondary Outcome: Change From Baseline in Health-related Quality of Life (HRQoL) as Assessed by EORTC-QLQ-C30 Score
Description: EORTC QLQ-C30 scale consists of 30 questions that assess participant functioning (physical, emotional, role, cognitive, and social), symptom (fatigue, nausea and vomiting, pain), global health/quality of life (QoL), and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Change in HRQoL was assessed using participant responses to questions regarding Global Health Status (Question 29: GHS; "How would you rate your overall health during the past week?") and QoL (Question 30: QoL; "How would you rate your overall quality of life during the past week?") were scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized. Scores range from 0-100. A higher score indicates a better outcome.
Time Frame: as for outcome 7
Population: ITT population included all randomized participants, regardless of whether they received any of the assigned treatment. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Atezolizumab
Number analyzed (Participants) | 198 | 200
score on a scale
  Baseline (Cycle 1 Day 1) | 66.92 (21.41) | 67.54 (20.79)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 192 | 192
  Change at Cycle 2 Day 1 | 2.99 (20.32) | 0.09 (18.33)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 190 | 187
  Change at Cycle 3 Day 1 | 4.87 (24.02) | 0.49 (17.35)
  Change at Cycle 4 Day 1: number analyzed (Participants) | 175 | 180
  Change at Cycle 4 Day 1 | 6.05 (21.04) | 1.34 (17.33)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 170 | 168
  Change at Cycle 5 Day 1 | 5.29 (22.80) | 1.19 (18.25)
  Change at Cycle 6 Day 1: number analyzed (Participants) | 168 | 163
  Change at Cycle 6 Day 1 | 4.66 (23.81) | 3.17 (18.01)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 161 | 155
  Change at Cycle 7 Day 1 | 7.25 (21.71) | 4.09 (17.47)
  Change at Cycle 8 Day 1: number analyzed (Participants) | 155 | 151
  Change at Cycle 8 Day 1 | 7.58 (21.48) | 4.25 (19.93)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 152 | 147
  Change at Cycle 9 Day 1 | 6.30 (23.20) | 3.00 (17.93)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 149 | 143
  Change at Cycle 10 Day 1 | 7.83 (22.29) | 3.85 (17.12)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 146 | 139
  Change at Cycle 11 Day 1 | 7.65 (21.21) | 2.64 (17.35)
  Change at Cycle 12 Day 1: number analyzed (Participants) | 145 | 138
  Change at Cycle 12 Day 1 | 7.47 (22.52) | 2.60 (17.75)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 140 | 136
  Change at Cycle 13 Day 1 | 8.45 (21.37) | 2.94 (18.41)
  Change at Cycle 14 Day 1: number analyzed (Participants) | 135 | 128
  Change at Cycle 14 Day 1 | 6.91 (21.82) | 3.39 (17.04)
  Change at Cycle 15 Day 1: number analyzed (Participants) | 134 | 125
  Change at Cycle 15 Day 1 | 7.21 (21.58) | 5.27 (18.13)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 123 | 117
  Change at Cycle 16 Day 1 | 6.30 (22.87) | 6.05 (17.83)
  Change at Study Discontinuation: number analyzed (Participants) | 179 | 177
  Change at Study Discontinuation | 3.86 (23.64) | 1.55 (18.41)
  Change at Follow Up 1: number analyzed (Participants) | 50 | 50
  Change at Follow Up 1 | 1.50 (25.01) | -5.83 (25.32)
  Change at Follow Up 2: number analyzed (Participants) | 41 | 44
  Change at Follow Up 2 | 4.67 (21.33) | -0.95 (21.73)
  Change at Follow Up 3: number analyzed (Participants) | 33 | 33
  Change at Follow Up 3 | -1.77 (18.84) | 2.53 (18.57)
  Change at Follow Up 4: number analyzed (Participants) | 34 | 28
  Change at Follow Up 4 | 0.74 (25.32) | 3.87 (22.51)
  Change at Follow Up 5: number analyzed (Participants) | 29 | 21
  Change at Follow Up 5 | 3.16 (23.19) | 4.76 (23.36)
  Change at Follow Up 6: number analyzed (Participants) | 29 | 18
  Change at Follow Up 6 | 6.32 (23.11) | 1.85 (17.28)
  Change at Follow Up 7: number analyzed (Participants) | 17 | 13
  Change at Follow Up 7 | 2.45 (23.34) | -10.26 (23.11)
  Change at Follow Up 8: number analyzed (Participants) | 17 | 11
  Change at Follow Up 8 | -8.33 (32.00) | 2.27 (11.84)
  Change at Follow Up 9: number analyzed (Participants) | 9 | 9
  Change at Follow Up 9 | 3.70 (17.24) | -1.85 (12.34)
  Change at Follow Up 10: number analyzed (Participants) | 5 | 8
  Change at Follow Up 10 | -15.00 (50.14) | 9.38 (9.38)
  Change at Follow Up 11: number analyzed (Participants) | 9 | 4
  Change at Follow Up 11 | -4.63 (50.88) | -4.17 (19.84)
  Change at Follow Up 12: number analyzed (Participants) | 5 | 4
  Change at Follow Up 12 | 20.00 (40.23) | -14.58 (20.83)
  Change at Follow Up 13: number analyzed (Participants) | 6 | 3
  Change at Follow Up 13 | 11.11 (38.61) | -2.78 (12.73)
  Change at Follow Up 14: number analyzed (Participants) | 2 | 1
  Change at Follow Up 14 | 8.33 (11.79) | -16.67 (0)
  Change at Follow Up 15: number analyzed (Participants) | 4 | 0
  Change at Follow Up 15 | 14.58 (34.94) |
  Change at Follow Up 16: number analyzed (Participants) | 3 | 0
  Change at Follow Up 16 | 2.78 (12.73) |
  Change at Follow Up 17: number analyzed (Participants) | 2 | 0
  Change at Follow Up 17 | -8.33 (11.79) |
  Change at Follow Up 18: number analyzed (Participants) | 2 | 0
  Change at Follow Up 18 | 8.33 (11.79) |

9. Secondary Outcome: Number of Participants With at Least One Adverse Event (AE)
Description: An AE is untoward medical occurrence in participant administered a pharmaceutical product & regardless of causal relationship with this treatment. An AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with use of investigational product, whether or not considered related to investigational product.
Time Frame: From first dose of study drug until 90 days after the last dose of study drug (up to 1 year, 3 months)
Population: Safety evaluable population included all randomized participants who received any amount of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Atezolizumab
Number analyzed (Participants) | 203 | 202
Participants | 186 | 192

10. Secondary Outcome: Serum Concentration of Atezolizumab
Time Frame: Predose and 0.5 hours post dose on Cycle 1 Day 1; Predose on Day 1 of Cycles 2, 4, 8, and 16 (Cycle length=21 days); study discontinuation visit (up to 1 year)
Population: Pharmacokinetic (PK)-evaluable population included all participants who received at least one dose of atezolizumab and provided at least one PK sample that was evaluable. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at specified timepoint. Different participants may have contributed data for each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliters (ug/mL)
Arm/Group | Atezolizumab
Number analyzed (Participants) | 194
micrograms per milliliters (ug/mL)
  Cycle 1 Day 1: Predose: number analyzed (Participants) | 187
  Cycle 1 Day 1: Predose | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not evaluable as samples were below lower limit of quantification (BLLQ).
  Cycle 1 Day 1: 0.5 hours Post-dose: number analyzed (Participants) | 183
  Cycle 1 Day 1: 0.5 hours Post-dose | 447 (27.1)
  Cycle 2 Day 1: Predose: number analyzed (Participants) | 191
  Cycle 2 Day 1: Predose | 99.2 (31.1)
  Cycle 4 Day 1: Predose: number analyzed (Participants) | 174
  Cycle 4 Day 1: Predose | 186 (64.3)
  Cycle 8 Day 1: Predose: number analyzed (Participants) | 137
  Cycle 8 Day 1: Predose | 238 (40.6)
  Cycle 16 Day 1: Predose: number analyzed (Participants) | 113
  Cycle 16 Day 1: Predose | 257 (40.3)
  Study Discontinuation: number analyzed (Participants) | 170
  Study Discontinuation | 178 (141.0)

11. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) to Atezolizumab
Description: Number of participants positive for Treatment Emergent ADA is the number of post-baseline evaluable participants determined to have treatment induced ADA or treatment-enhanced ADA during the study period.
Time Frame: Predose on Day 1 of Cycles 1, 2, 4, 8 and 16 (Cycle length=21 days)
Population: ADA evaluable population included all randomized participants who received at least one dose of atezolizumab and who had at least one post-baseline ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 192
Participants | 13

ADVERSE EVENTS:
Time Frame: For adverse events (AEs): From first dose of study drug until 90 days after the last dose of study drug (up to 1 year, 3 months); For all-cause mortality: from randomization through the end of post-treatment survival follow-up (up to 5 years, 5 months)
Description: Safety-evaluable population included all randomized participants who received any amount of the study treatment.
Arm/Group | Placebo | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 69/203 | 70/202
Serious Adverse Events (participants affected / at risk) | 32/203 | 32/202
Other Adverse Events (participants affected / at risk) | 144/203 | 155/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=203) | Atezolizumab (N=202)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 2 (2)
Implant site pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (3) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pericoronitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngolaryngeal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 6 (6)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative adhesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal necrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fistula repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastrostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Medical device removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Muscle flap operation (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=203) | Atezolizumab (N=202)
Anaemia (Blood and lymphatic system disorders) | 18 (21) | 19 (24)
Lymphopenia (Blood and lymphatic system disorders) | 22 (36) | 8 (11)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 11 (11)
Hypothyroidism (Endocrine disorders) | 34 (36) | 54 (59)
Constipation (Gastrointestinal disorders) | 5 (5) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 26 (40)
Dry mouth (Gastrointestinal disorders) | 16 (16) | 18 (21)
Asthenia (General disorders) | 16 (22) | 11 (20)
Fatigue (General disorders) | 26 (30) | 29 (32)
Alanine aminotransferase increased (Investigations) | 5 (8) | 13 (17)
Aspartate aminotransferase increased (Investigations) | 6 (10) | 12 (14)
Blood creatinine increased (Investigations) | 7 (7) | 11 (16)
Weight decreased (Investigations) | 11 (11) | 13 (15)
Decreased appetite (Metabolism and nutrition disorders) | 16 (16) | 16 (17)
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 (17) | 6 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (22) | 22 (27)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 12 (13)
Headache (Nervous system disorders) | 11 (11) | 14 (22)
Anxiety (Psychiatric disorders) | 5 (5) | 12 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 17 (21)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 6 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (17) | 23 (27)
Rash (Skin and subcutaneous tissue disorders) | 17 (18) | 13 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT03452137/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT03452137/SAP_001.pdf